CLINICAL TRIAL: NCT02858505
Title: Impact of One Versus Two Amino Acid Chelated Iron Capsules on Prevention of Iron Deficiency Anemia in Non-anemic Women With Twin Gestations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IDAT
Record Dates: First submitted 2016-08-02; First posted 2016-08-08 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 27 mg elemental iron group (Active Comparator): received 27 mg elemental iron once daily starting at 12 weeks until 36 weeks
  Interventions: Drug: 27 mg elemental iron
- 54 mg elemental iron group (Active Comparator): received 54 mg elemental iron once daily starting at 12 weeks until 36 weeks
  Interventions: Drug: 54 mg elemental iron

INTERVENTIONS:
Drug: 27 mg elemental iron
  Arms: 27 mg elemental iron group
Drug: 54 mg elemental iron
  Arms: 54 mg elemental iron group

SUMMARY:
Anaemia is the most worldwide health problem affecting pregnant women in both developed and developing countries. During pregnancy there is an inconsistent increase in plasma volume and haemoglobin mass.

Iron deficiency anemia is the commonest type of anemia during pregnancy. The pregnant woman needs about 1000 mg of iron during pregnancy.

Diet alone cannot give pregnant woman the daily required amount of the iron (about 27 mg/day) so the Centers for Disease Control and Prevention recommend that pregnant women take a daily supplement of 30 mg of elemental iron as a preventive dose. As most women begin their pregnancy with low iron stores, particularly in the second and third trimesters, so prevention should start as soon as possible even before pregnancy to prevent depletion of iron store and further Iron deficiency anemia.

Oral iron is a cheap, effective and relatively safe line to prevent Iron deficiency anemia during pregnancy. The common available ferrous salts include ferrous fumarate, ferrous sulphate and ferrous gluconate. Unfortunately; these iron forms are associated usually with constipation, darkened stools, diarrhea, loss of appetite, nausea, stomach cramps, and vomiting.

Iron amino acid chelates have been emerged to be used as agents for prevention and treatment of Iron deficiency anemia. These agents provide maximum bioavailability and maximum efficacy with minimal unpleasant side effects.

Twin pregnancies have a significant role in perinatal morbidity due to increased risks of low birth weight and preterm birth. The iron requirement for twin pregnancy is probable double fold that of a singleton pregnancy and maternal hemoglobin in twin gestations is usually lower than in singleton pregnancy resulting in higher rate of Iron deficiency anemia.

ELIGIBILITY:
Inclusion Criteria:

* twin gestations
* ±12 weeks)
* normal hemoglobin level (Hb ≥ 120 g/L).
* women were living in nearby area to make up follow up quit possible
* willing to participate in our study

Exclusion Criteria:

* a recent blood transfusion
* threatened miscarriage
* pathological blood loss
* vegetarian diet
* intolerant to oral iron form
* history of haematologic disorder
* chronic diseases
* unwillingness to co-operate.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2015-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Hemoglobin level | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes